CLINICAL TRIAL: NCT07392346
Title: A Prospective, Single-Arm, Phase Ⅱ Clinical Trial Evaluating Fruquintinib in Combination With Paclitaxel for Injection (Albumin-bound) and Iparomlimab and Tuvonralimab Injection as Second-Line Therapy in Advanced Gastric Cancer Patients Previously Received Immunotherapy
Brief Title: Safety and Efficacy of Fruquintinib Plus Nab-Paclitaxel and Iparomlimab and Tuvonralimab Injection in the Second-Line Treatment for Immunotherapy-experienced Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dai, Guanghai (Other)
Responsible Party: Sponsor-Investigator, Dai, Guanghai, Professor,Chief Physician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2026-003
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Gastric Cancer Adenocarcinoma Metastatic
MeSH Terms: interventions — HMPL-013; Taxes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Fruquintinib Plus Nab-Paclitaxel and Iparomlimab and Tuvonralimab Injection are administered until disease progression or toxicity intolerable.
  Interventions: Drug: Fruquintinib; Drug: Iparomlimab and Tuvonralimab; Drug: Paclitaxel (albumin-bound)

INTERVENTIONS:
Drug: Fruquintinib — 3 mg qd, po, q3W; After 6 cycles of combination therapy, maintenance treatment consisting of Iparomlimab and Tuvonralimab Injection plus Fruquintinib will continue until disease progression, intolerable toxicity, initiation of new antitumor therapy, withdrawal of informed consent, or investigator's determination that the subject should discontinue from study treatment.
Drug: Iparomlimab and Tuvonralimab — 5.0 mg/kg, Day 1, q3W, iv. After 6 cycles of combination therapy, maintenance treatment consisting of Iparomlimab and Tuvonralimab Injection plus Fruquintinib will continue until disease progression, intolerable toxicity, initiation of new antitumor therapy, withdrawal of informed consent, or investigator's determination that the subject should discontinue from study treatment.
Drug: Paclitaxel (albumin-bound) — 250 mg/m², Day 1, q3W

SUMMARY:
Immunotherapy has established the new standard for first-line treatment of advanced or metastatic gastric cancer. However, current second-line options-predominantly consisting of targeted therapy plus chemotherapy or chemotherapy alone-confer only modest clinical benefit. Notably, pivotal phase III second-line trials (REGARD, RAINBOW, RAINBOW-Asia, FRUTIGA) exclusively enrolled patients who progressed on chemotherapy regimens; thus, high-quality evidence guiding second-line treatment specifically for immunotherapy-refractory patients remains scarce, representing a significant unmet medical need.

Anti-angiogenic agents have demonstrated capacity to ameliorate the hypoxic, immunosuppressive tumor microenvironment while exerting synergistic anti-tumor effects when combined with immune checkpoint inhibitors. Exploratory studies evaluating immunotherapy combined with anti-angiogenic therapy plus chemotherapy in advanced gastric cancer patients after first-line failure have yielded encouraging efficacy signals (NCT03966118, NCT04982276), with objective response rates of 30-40% and median progression-free survival approaching 6 months.

Based on this, the investigators aim to evaluate the efficacy and safety profile of fruquintinib combined with nab-paclitaxel and Iparomlimab and Tuvonralimab Injection (a novel bispecific antibody) as second-line treatment for patients with advanced gastric cancer who have experienced disease progression during or after first-line immunotherapy-containing regimens.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years
2. Pathologically or cytologically confirmed diagnosis of gastric cancer (GC) or gastroesophageal junction (GEJ) cancer.
3. Failure of first-line treatment with PD-1/PD-L1 inhibitors
4. With measurable lesions according to RECIST 1.1 criteria.
5. ECOG performance status of 0-1
6. Expected survival ≥3 months;
7. Major organ functions meet the following requirements :

   * Absolute neutrophil count (ANC) ≥ 1,500/mm³ (1.5 × 10⁹/L) (no growth factors used within 14 days).
   * Platelet count (PLT) ≥ 100,000/mm³ (100 × 10⁹/L) (no correction therapy used within 7 days).
   * Hemoglobin (Hb) ≥ 9 g/dL (90 g/L) (no correction therapy used within 7 days).
   * Serum creatinine ≤ 1.5 × upper limit of normal (ULN).
   * Total bilirubin (BIL) ≤ 1.5 × upper limit of normal (ULN).
   * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) levels ≤ 2.5 × upper limit of normal (ULN); ≤ 5 × upper limit of normal (ULN) for patients with liver metastases.
   * Urinalysis is normal, or urine protein < (++), or 24-hour urine protein level < 1.0 g.
8. Normal coagulation function, with no history of active bleeding or thrombotic diseases:

   * International normalized ratio (INR) ≤ 1.5 × ULN.
   * Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
   * Prothrombin time (PT) ≤ 1.5 × ULN.
9. For patients with potential fertility, the following requirements must be met:

   * Adopt a medically acceptable contraceptive method (e.g., intrauterine device, oral contraceptives, or condoms) during the study treatment period and for 3 months after the completion of study treatment.
   * Serum human chorionic gonadotropin (β-HCG) test must be negative within 72 hours prior to study enrollment.
   * Must not be breastfeeding.
10. Patients must have provided written informed consent, and be willing and able to comply with the scheduled visits, study treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. History of gastrointestinal perforation and/or fistula within 6 months prior to the first dose of study medication.
2. Uncontrolled pleural, pericardial, or peritoneal effusions requiring repeated drainage.
3. Hypersensitivity to any component of monoclonal antibodies, fruquintinib, or albumin-bound paclitaxel.
4. Receipt of any of the following treatments:

   1. Severe adverse reactions to prior immunotherapy.
   2. Prior treatment with CTLA4 inhibitors.
   3. Any study medication within 4 weeks prior to the first dose of study medication.
   4. Concurrent enrollment in another clinical study (excluding observational studies or survival follow-ups of interventional studies).
   5. Last dose of anti-cancer therapy ≤ 3 weeks prior to the first study medication, or fixed-field palliative radiotherapy ≤ 2 weeks prior to study intervention.
   6. Corticosteroid use (>10 mg prednisone equivalent/day) within 2 weeks prior to study medication; the investigator may decide on eligibility in special cases. Inhaled/topical steroids and adrenal replacement at >10 mg/day prednisone equivalent are permitted in the absence of active autoimmune diseases.
   7. Anti-tumor vaccines or live vaccines within 4 weeks prior to study medication.
   8. Major surgery or severe trauma within 4 weeks prior to study medication.
5. Previous anti-tumor treatment toxicities not recovered to ≤ CTCAE Grade 1 (excluding alopecia) or the specified inclusion/exclusion criteria levels.
6. Central nervous system metastases.
7. History of active autoimmune diseases (e.g., interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism) or a history of such diseases (excluding vitiligo, or childhood asthma/allergies cured and requiring no intervention in adulthood; autoimmune hypothyroidism on stable thyroid replacement; type 1 diabetes on stable insulin).
8. Immunodeficiency history (including HIV-positive status, acquired/congenital immunodeficiency, organ transplantation, or allogeneic bone marrow transplantation).
9. Inadequately controlled cardiovascular symptoms/diseases, including: (1) NYHA Class II or higher heart failure; (2) Unstable angina; (3) Myocardial infarction within 1 year; (4) Clinically significant supraventricular/ventricular arrhythmias (uncontrolled with clinical intervention).
10. Urinalysis showing urine protein ≥++ and confirmed 24-hour urine protein >1.0 g.
11. Abnormal coagulation (INR >1.5×ULN or PT >ULN+4s), with bleeding tendency or thrombolytic/anticoagulant therapy (small-dose low-molecular-weight heparin or oral aspirin for prophylaxis permitted during the trial).
12. Significant clinical bleeding or definite bleeding tendency within 3 months (e.g., gastrointestinal bleeding, hemorrhagic gastric ulcer, vasculitis). If baseline occult blood in stool is positive, re-testing is allowed; endoscopy may be performed based on clinical judgment if positive after re-testing.
13. Active ulcers, unhealed wounds, or fractures.
14. Hypertension inadequately controlled by anti-hypertensive medication (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg).
15. Severe infection (CTCAE >Grade 2) within 4 weeks prior to study medication (e.g., severe pneumonia, bacteremia, infectious complications requiring hospitalization); baseline chest imaging showing active pulmonary inflammation, or infection symptoms/signs requiring oral/IV antibiotics within 2 weeks prior to study medication (excluding prophylactic antibiotics).
16. History of interstitial lung disease (excluding radiation pneumonitis or non-infectious pneumonitis not treated with steroids).
17. Active tuberculosis (confirmed by history/CT) or history of active tuberculosis within 1 year prior to enrollment, or untreated active tuberculosis more than 1 year prior to enrollment.
18. History of any other malignant tumor within 5 years prior to study medication (excluding low-risk tumors with >90% 5-year survival rate, e.g., adequately treated basal cell/squamous cell skin cancer or cervical intraepithelial neoplasia).
19. Pregnant or breastfeeding women.
20. Other factors (e.g., concurrent severe diseases including mental illness, severely abnormal lab values, family/social factors) that may lead to forced withdrawal from the study, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Progress-free Survival(PFS) | 24 months
  The time from enrollment until tumor progression or death from any cause, whichever occurred first

SECONDARY OUTCOMES:
Objective response rate (ORR) | 24 months
  The proportion of patients with a confirmed complete response or partial response
Disease control rate (DCR) | 24 months
  The proportion of patients with a best overall response of confirmed complete or partial response, or stable disease
Overall Survival (OS) | 24 months
  The time from randomization to death from any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided